CLINICAL TRIAL: NCT07212140
Title: Adaptation of the STAIR-NT Intervention to Respond to Psychological Health Conditions for First Responders With a History of Traumatic Brain Injury
Brief Title: Adaptation of the STAIR-NT for First Responders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Invisible Wounds Project (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joseph Schwartz, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005143; HT9425-24-1-0782 (Other Grant/Funding Number: Department of Defense (DOD))
Record Dates: First submitted 2025-09-25; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-02

CONDITIONS: PTSD - Post Traumatic Stress Disorder; TBI-Traumatic Brain Injury
Keywords: PTSD; TBI; First responders; STAIR-NT; GMT
MeSH Terms: conditions — Combat Disorders; Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic | interventions — Narrative Therapy

STUDY DESIGN:
Intervention Model Description: Pilot randomized control trial with an intervention arm and a treatment-as-usual arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted STAIR-NT Intervention (Experimental): Participants in this arm will receive the adapted version of Skills Training in Affective and Interpersonal Regulation-Narrative Therapy (STAIR-NT).
  Interventions: Behavioral: Adapted STAIR-NT
- Treatment as usual (TAU) (No Intervention): Participants in this arm will receive treatment as usual.

INTERVENTIONS:
Behavioral: Adapted STAIR-NT — An adapted version of STAIR-NT that utilizes components from GMT in order to treat PTSD and TBI.
  Other Names: Skills Training in Affective and Interpersonal Regulation with Narrative Therapy
  Arms: Adapted STAIR-NT Intervention

SUMMARY:
This study is a randomized controlled pilot examining the implementation of an adapted intervention, Skills Training in Affective and Interpersonal Regulation-Narrative Therapy (STAIR-NT), among a first responder population with a history of TBI and PTSD.

DETAILED DESCRIPTION:
The primary objective of the study is to implement and evaluate the effectiveness of an evidence-based intervention, STAIR-NT, which will be adapted with Goal Management Training (GMT). A small-scale randomized control pilot will be conducted using the adapted intervention to examine implementation (i.e., feasibility, acceptability) and improvements in short-term PTSD, as well as secondary mental health outcomes (e.g., anxiety, and depression symptoms, substance misuse) among a first responder population with a history of TBI and PTSD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* be a first responder within the state of Minnesota
* have a history of a TBI
* screen for PTSD.

Exclusion Criteria:

* Does not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Post-Traumatic Stress Disorder Symptoms | Baseline, 4-6 weeks, 3 months, 6 months
  The 20-item PTSD Checklist for DSM-5 (PCL-5) will be used to assess PTSD symptoms. All items are scored on a 5-point Likert scale ranging between 0 (not at all) and 4 (extremely).

SECONDARY OUTCOMES:
Change in Anxiety Symptoms | Baseline, 4-6 weeks, 3 months, 6 months
  The Generalized Anxiety Disorder Screener-7 (GAD-7) will be used to assess anxiety symptoms. The included items ask participants to indicate how frequently they experienced seven symptoms over the past two weeks, with provided response categories ranging between 0 (not at all) to 3 (nearly every day).
Change in Depression Symptoms | Baseline, 4-6 weeks, 3 months, 6 months
  The Patient Health Questionnarie-9 (PHQ-9) is an abbreviated version of the full PHQ focused on major depressive disorder and will be used to assess depression symptoms. Participants are asked to indicate how often they experienced nine different feelings over the past two weeks with possible response categories ranging between 0 (not at all) and 3 (nearly every day).
Change in Alcohol Use | Baseline, 4-6 weeks, 3 months, 6 months
  The Alcohol Use Disorders Identification Test (AUDIT) is a self-administered instrument that includes 10 screening questions tapping alcohol use and alcohol-related consequences in the past 12 months.
Change in Drug Use | Baseline, 4-6 weeks, 3 months, 6 months
  The Drug Abuse Screening Test (DAST-10) is a 10-item questionnaire tapping the use of drugs and related health effects and behaviors over the past 12 months.

OTHER OUTCOMES:
Change in General Well Being | Baseline, 4-6 weeks, 3 months, 6 months
  The General Well Being Schedule (GWB) is an 18-item, self-administered questionnaire that includes positive and negative questions tapping six dimensions: positive well-being, self-control, vitality, depression, anxiety, and general health. Statements ask participants to indicate feelings in the past 30 days. Lower scores indicate lower overall well-being.
Changes in Health Conditions | Baseline, 4-6 weeks, 3 months, 6 months
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a 12-item questionnaire tapping difficulties due to health conditions. Participants report difficulties in physical, cognitive, and social tasks in the past 30 days. Provided response categories range between 0 (none) and 4 (extreme or cannot do).
Change in Social Support | Baseline, 4-6 weeks, 3 months, 6 months
  The Medical Outcomes Study (MOS) Social Support Survey is a 19-item self-administered questionnaire tapping four functional support domains: positive social interaction, emotional/informational support; tangible/instrumental support; and affectionate support. Provided response categories range from "none of the time" to "all of the time"
Changes in Chronic Pain | Baseline, 4-6 weeks, 3 months, 6 months
  The Brief Pain Inventory-Short Form (BPI-SF), is a 15-item self-administered questionnaire that assesses the severity and impact of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Schwartz, PhD, Principal Investigator — Florida State University
Locations (1):
- Invisible Wounds Project, Forest Lake, Minnesota, United States